CLINICAL TRIAL: NCT00837837
Title: A Single-Dose, Open-Label, Pharmacokinetic Study of Chlorpheniramine Maleate Liquid in Children and Adolescents
Brief Title: Study Evaluating Chlorpheniramine Maleate Liquid in Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-08-01
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Allergic Reactions
Keywords: pharmacokinetics; children; adolescents; antihistamine
MeSH Terms: conditions — Hypersensitivity | interventions — Chlorpheniramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chlorpheniramine (Experimental): Chlorpheniramine dose by body weight.
  Interventions: Drug: Chlorpheniramine

INTERVENTIONS:
Drug: Chlorpheniramine

SUMMARY:
The purpose of this study is to examine the pharmacokinetic parameters of chlorpheniramine in children and adolescents.

DETAILED DESCRIPTION:
This is a single-group, single-center, open-label, one period, bioavailability study. This study will evaluate the pharmacokinetic (PK) profile of chlorpheniramine in a population of children aged 2 to <12 yrs and adolescents aged 12 to <18 yrs. Twelve blood samples (3.0 mL) for chlorpheniramine analysis will be drawn at time 0 (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours after dosing. Plasma levels of chlorpheniramine will be determined. The following primary, single-dose PK parameters for chlorpheniramine will be determined using noncompartmental methods: AUCL, AUCI, and Cmax. The following PK parameters will also be determined to provide a complete profile of the drug, as appropriate: oral clearance (CL) and volume of distribution (Vd) and adjusted for body weight (per kg); time to reach Cmax (tmax), and apparent elimination constant (Kel) and half-life (t1/2). The PK parameters will be summarized using descriptive statistics.

ELIGIBILITY:
INCLUSION CRITERIA:

Individuals may be enrolled in the study if they meet all of the following criteria:

1. Males or females between 2 to <18 yrs of age with a minimum weight of 24 pounds and within the 5th and 95th percentiles in physical growth characteristics (i.e., height and weight) and BMI based on age and gender,
2. Symptomatic or asymptomatic children/adolescents as follows:

i.A prior diagnosis of allergic rhinitis and either symptomatic or asymptomatic at the time of entry in the study; or ii.Symptoms of an acute Upper Respiratory Infection (URI); or iii.No symptoms of an acute URI, but at risk for developing an acute URI as evidenced by the following frequency, crowding, and exposure criteria:

* Frequency: a history of frequent URIs defined as >6 infections/yr for children aged 2 to <6 yrs and as >4 infections per year for adolescents aged 6 to <18 yrs;
* Crowding: living in a home with ≥4 persons, or sleeping in the same bedroom with ≥3 persons;
* Exposure: the presence of another family member in the household who is ill with a URI, or a child in the family that is attending preschool, or attending school with ≥6 children in the class; c.Except for allergic rhinitis or a URI, children/adolescents are in normal physical health (i.e., no clinically significant systemic disease) as judged by the Investigator upon physical examination of the subject; d.Subjects do not require concomitant medication except for low-dose inhaled glucocorticoids for allergic rhinitis or mild concomitant asthma, if dose is stabilized before entry in the study (i.e., dose is not changed for one month prior to or during the study), and inhaled short-acting beta-2 adrenergic agonists for concomitant asthma, as needed; e.Post menarchal females must be using a reliable method of contraception (i.e., oral, transdermal, injectable or implanted contraceptives, IUD, cervical cap, diaphragm, condom, abstinence, or surgical sterility); f.Parent/guardian/adolescent provides written informed consent and child provides assent, if age appropriate.

EXCLUSION CRITERIA:

Individuals are not eligible for entry in the study if any of the following are noted:

1. The child/adolescent weighs <24 pounds or is below the 5th or above the 95th percentiles in physical growth characteristics (i.e., height and weight) and BMI based on age and gender;
2. Inability to swallow the medication;
3. Eaten within 2 hours prior to dosing;
4. A known hypersensitivity to CHLOR, any other antihistamine, or EMLA® cream;
5. Systolic and/or diastolic blood pressure at or above the 95th percentile based on gender, and age and height percentiles. (Note: If a subject with no history of hypertension has a blood pressure reading at or above the 95th percentile, the subject will be allowed to rest for 15 minutes and the blood pressure measurement repeated. Up to 3 consecutive measurements at approximately 5 min intervals will be allowed. Subjects who continue to have systolic and/or diastolic blood pressure readings at or above the 95th percentile will be excluded from the study);
6. History of melena or any hepatic, renal, endocrine (e.g., diabetes, thyroid disorder), cardiac, neurological, psychiatric, gastrointestinal, hematological or metabolic disorder deemed to be clinically significant by the Investigator;
7. Any serious medical condition or medical history felt by the Investigator to place them at increased risk;
8. The child is diagnosed with anemia or has a red blood cell count or hemoglobin level outside of normal range as evidenced by baseline hematology assessment;
9. Asthma symptoms at the time of entry in the study or requires medication other than allowed under Inclusion Criterion d;
10. Failure to comply with appropriate washout periods for any H-1 receptor antagonist treatment before and during the study, i.e., no use within 7 days of entering the study or at any time during the study, and no use of astemizole within the preceding 3 calendar months;
11. Other than described in Exclusion Criterion i, use of any medication 72 hours prior to dosing;
12. A history of drug, alcohol, or tobacco abuse (older children and adolescents), a history of Hepatitis B, a previous positive test for Hepatitis B surface antigen, or a previous positive Hepatitis C antibody;
13. A history of HIV infection or previous demonstration of HIV antibodies;
14. Female subjects who have experienced menarche and have a positive urine pregnancy test;
15. Parent/guardian/subject judged by the Investigator to be unable or unwilling to comply with the requirements of the protocol;
16. Have taken an investigational drug within 30 days prior to entering the study or have already participated in the trial;
17. Relative of the Sponsor, Investigator, or any personnel of the study site who are directly involved with the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2008-12-21 (Actual); Primary Completion 2009-02-02 (Actual); Study Completion 2009-02-02 (Actual)

PRIMARY OUTCOMES:
AUC and Cmax | 72 hours

SECONDARY OUTCOMES:
Oral clearance (CL) and volume of distribution (Vd); time to reach Cmax (tmax), and apparent elimination constant (Kel) and half-life (t1/2). | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Pathirana S, Jayawardena S, Meeves S, Thompson GA. Brompheniramine and Chlorpheniramine Pharmacokinetics Following Single-Dose Oral Administration in Children Aged 2 to 17 Years. J Clin Pharmacol. 2018 Apr;58(4):494-503. doi: 10.1002/jcph.1037. Epub 2017 Nov 14. PMID 29136286